CLINICAL TRIAL: NCT05996367
Title: Prospective Cohort Assessing the Impact of Single-dose Radiotherapy in the Treatment of Painful Bone Lesions in Patients With Multiple Myeloma
Brief Title: Prospective Cohort of Single-dose Radiotherapy for Painful Bone Lesions in Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Geovanne Pedro Mauro, Primary Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 465/23
Record Dates: First submitted 2023-07-31; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Palliative care; Radiotherapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single-dose radiation to involved-site
  Interventions: Radiation: Single-dose involved-site radiotherapy

INTERVENTIONS:
Radiation: Single-dose involved-site radiotherapy — Single-dose of 8 Gy at involved-site radiotherapy

SUMMARY:
Multiple myeloma is a plasma cell neoplasm that can cause painful bone lesions. The main treatment for these lesions and pain control is radiotherapy, usually in daily fractions. In 2017, a phase III study proved the effectiveness of using a single dose of 8 Gy, but without description of several important oncological outcomes. This is a single-arm prospective cohort study. This study aims to describe these outcomes, including retreatment rate and bone events. Also, as secondary objectives, describe the quality of life and use of analgesic medications in this population.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy of plasma cell neoplasm with bone lesion treatable with radiotherapy;
* Age between 18 and 85 years old;
* Performance on the ECOG scale less than or equal to 2.
* Not using systemic therapies for 4 weeks OR being on maintenance therapy with the same drug for at least 4 weeks before radiotherapy.

Exclusion Criteria:

* Refusing to sign or inability to understand the consent term;
* Pain less than 2/10 on the numeric pain rating scale;
* Change in systemic treatment scheme, including use of bone metabolism modulation drugs, up to 4 weeks before radiotherapy treatment;
* Technical incapacity for the treatment, including, but not limited to, weight greater than 115Kg, inability to abduct the limb to be treated in appendicular bones, intolerable pain to remain in the treatment position;
* Previous cancer and previous oncological treatments;
* Previous autoimmune diseases, even if controlled;
* Current pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Retreatment rate at 6 months | 6 months after radiotherapy
  Percentage of patients that needed a second corse of radiation for painful bone lesions

SECONDARY OUTCOMES:
Local control | 6 months and 12 months
  Local control by Recist 1.1
Progression-free survival | 12 months
  Progression-free survival
Overall survival | 12 months
  Overall survival
Bone event-free survival | 6 months
  by description from Raje et al. The Lancet 2018
Pain relief by the numerical rating pain scale | 1, 3, 6 and 12 months
  reduction on opioid and single analgesics intake and altered value in the rating pain scale
Pain flair incidence | 1, 3, 6 and 12 months
  Enhanced pain by at least 2 levels at the numerical rating pain scale
Quality of life by EORCT QLQ-C30 | 1, 6 and 12 months
  Quality of life by EORCT QLQ-C30 questionnaire
Quality of life by EORCT QLQ-C30 and MY-24 | 1, 6 and 12 months
  Quality of life by EORCT MY-24 myeloma complementary questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Geovanne P Mauro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No